CLINICAL TRIAL: NCT04190238
Title: Efficiency of the Super Inductive System in Spasticity Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Ciubean Alina Deniza, Principal investigator, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversitateaMFHCJ
Record Dates: First submitted 2019-12-02; First posted 2019-12-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Spasticity, Muscle
MeSH Terms: conditions — Muscle Spasticity | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: case-control study
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spasticity after stroke 1 (Experimental): Physical therapy with super inductive system on the agonist and antagonist muscles
  Interventions: Other: Super inductive system (high frequency electromagnetic field); Other: Physical therapy
- Spasticity after stroke 2 (Active Comparator): Physical therapy with super inductive system on the antagonist muscles
  Interventions: Other: Super inductive system (high frequency electromagnetic field); Other: Physical therapy

INTERVENTIONS:
Other: Super inductive system (high frequency electromagnetic field) — Super inductive system (high frequency electromagnetic field)
Other: Physical therapy — specific for spasticity

SUMMARY:
The aim of the study is to see whether a physical therapy program can relieve pain, decrease spasticity and increase muscle contraction force by using the super inductive system (high frequency electromagnetic field). It is a longitudinal, prospective study, of 60 patients with spasticity after stroke. No new treatment method is tested, as the Super inductive system is approved for physical therapy by the Ministry of Health.

DETAILED DESCRIPTION:
The 60 patients will be submitted to 2 treatment groups: 30 patients will receive 10 sessions of the superinductive system on the antagonist muscles, and 30 patients will receive 10 sessions the superinductive system on the agonist and antagonist muscles. All patients will also receive the standard kinetotherapy program for spasticity. The patients will be evaluated at the beginning of the treatment, at 10 days and at 30 days by using the functional MAS index and Barthel index.

ELIGIBILITY:
Inclusion Criteria:

* spasticity after stroke

Exclusion Criteria:

* spasticity of other causes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
change in MAS functional index | day 0, day 10, day 30
  upper extremity functional index
change in Barthel index | day 0, day 10, day 30
  measurement of activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Viorela M Ciortea, MD, PhD, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu
Locations (1):
- Clinical Rehabilitation Hospital, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
if solicited
Supporting Information: Study Protocol
Time Frame: at the end of the study
Access Criteria: on demand by e-mail